CLINICAL TRIAL: NCT03030118
Title: Study of Anti-Malarials in Incomplete Lupus Erythematosus
Acronym: SMILE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Nancy Olsen, Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00003506; U01AR071077 (NIH)
Record Dates: First submitted 2017-01-15; First posted 2017-01-24 (Estimated); Results first posted 2025-08-29 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: hydroxychloroquine
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (Active Comparator): Hydroxychloroquine will be administered as a once daily dose of 200 or 400 mg, based on the patient's weight. Treatment will be for 96 weeks.
  Interventions: Drug: Hydroxychloroquine
- Placebo oral capsule (Placebo Comparator): Placebo will be administered as one or two capsules as a single daily dose, based on the patient's weight. Treatment will be for 96 weeks.
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine is classified as an anti-malarial and it is has immunomodulatory functions that make it useful for treatment of autoimmune disorders including systemic lupus erythematosus and rheumatoid arthritis.
  Other Names: Plaquenil
  Arms: Hydroxychloroquine
Drug: Placebo Oral Capsule — An oral capsule placebo is made to match the active intervention medication hydroxychloroquine.
  Other Names: Placebo
  Arms: Placebo oral capsule

SUMMARY:
This project is a multicenter, randomized, placebo-controlled, double-blind clinical trial that is designed to test whether treating patients who are at risk for development of lupus with hydroxychloroquine can slow accumulation of disease features. Effects on clinical progression of symptoms, patient-reported outcomes and changes in the immune markers of response will be measured and toxicity of the treatment will be assessed. This trial is a first step in testing a prevention strategy for lupus.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) causes major organ damage and shortens lifespan in relatively young persons. Early diagnosis and treatment are essential to improving outcomes for SLE patients. However, evidenced-based approaches to early treatment interventions and the appropriate target population for these interventions are not available. We propose that individuals who have positivity for antinuclear antibodies (ANAs) and who also exhibit some of the other features that are used to classify SLE, are at high risk of progressing to the full systemic form of this disease. These individuals, who have significant levels of ANA with 1 or 2 additional items from the lupus classification criteria, are considered to have incomplete lupus erythematosus (ILE). We propose to treat ILE patients with hydroxychloroquine (HCQ) in the "Study of Anti-Malarials in Incomplete Lupus Erythematosus" or SMILE trial. The primary objective is to determine whether HCQ treatment can prevent acquisition of additional clinical and immunologic features that define SLE.

The major secondary objectives are to determine whether HCQ treatment: (1) lessens lupus disease activity as measured by standard scoring indices; (2) improves patient reported outcomes (3) prevents accumulation of immunologic abnormalities including autoantibodies and cytokines and (4) has an acceptable toxicity profile. The specific aims of this proposal are:

1. To carry out a double-blind, placebo-controlled, multicenter, randomized trial of HCQ vs. placebo in patients with ILE. The study tests the hypothesis that early use of HCQ can modify disease features so that accumulation of abnormalities leading to a classification of SLE can be significantly slowed.
2. To determine effects of HCQ on disease activity and patient-reported outcomes in patients with ILE.
3. To characterize the immunologic profile of HCQ in ILE-treated patients. Autoantibodies, cytokines and chemokines will be measured on multiplex arrays for developing insights into underlying mechanisms.
4. To quantitatively assess the incidence of ophthalmologic toxicity in HCQ-treated ILE patients. All enrolled patients will have standardized ophthalmologic examinations before and after study treatment. Recommendations for use and monitoring in this patient population will be developed.

The SMILE trial will determine whether or not HCQ should be given to ILE patients, will provide insights into the appropriate target population, and will propose candidate biomarkers to guide treatment decisions. While not part of the Precision Medicine Initiative®, SMILE is consistent with its goals. It will be the first step towards testing the feasibility of disease prevention studies in SLE and will accumulate biological samples in a repository that will be available to the lupus research community for further in-depth mechanistic studies.

ELIGIBILITY:
Inclusion Criteria:

1. Between 15 and 49 years of age, inclusive, at Visit 1.
2. Anti-nuclear antibody (ANA) titer of 1:80, or greater, as determined by immunofluorescence assay (IFA).
3. Participants must have at least one (but not three or more) additional clinical or laboratory criterion from the 2012 Systemic Lupus International Collaborating Clinics (SLICC) classification criteria.
4. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. The subject meets the 2012 SLICC classification criteria for SLE at Visit 1 (i.e., ANA plus 3 other criteria, or ANA plus biopsy-proven lupus nephritis).
2. The subject has been diagnosed with another autoimmune disorder, other than autoimmune thyroid conditions.
3. The subject has fibromyalgia, based on clinical history and exam.
4. The subject has previously been or is currently being treated with oral antimalarial agents including hydroxychloroquine, chloroquine, or quinacrine.
5. The subject is currently or has been treated with immunosuppressive, immune modifying, or cytotoxic medications as listed in Section 7.2.
6. Use of any investigational agent within the preceding 12 months.
7. History of primary immunodeficiency.
8. Active bacterial, viral, fungal, or opportunistic infection.
9. Evidence of infection with human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C.
10. Concomitant malignancy or history of malignancy with the exception of adequately treated basal or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix.
11. The subject has significant findings on ophthalmological examination that, in the opinion of the examining Ophthalmologist, prevent safe use of hydroxychloroquine.
12. The subject has other contraindications to treatment with hydroxychloroquine including pre-existing ocular disease, hepatic impairment, psoriasis, porphyria, or allergy to the drug or class.
13. Co-morbidities requiring systemic corticosteroid therapy greater than 10 mg of prednisone per day, or equivalent, or a change in corticosteroid dose within the 3 months prior to Visit 1.
14. Starting, stopping, or changing the dose of over the counter or prescription non-steroidal anti-inflammatory drugs (NSAIDs) in the three months prior to Visit 1.
15. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
16. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
17. Inability to comply with the study visit schedule and procedures.

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 187 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Olsen, MD, Principal Investigator — Penn State MS Hershey Medical Center; David R Karp, MD PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (7):
- United States (7):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Northwell Health, Great Neck, New York
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Penn State MS Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other investigators upon reasonable request. This will include all patient-level measurements and instruments, as well as the laboratory results.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after publication of the primary paper, anticipated in last quarter 2025.
Access Criteria: Reasonable request is defined as having a legitimate and specific purpose for use of the data and ability to accept it in a usable format.

REFERENCES:
- [Background] Karp DR, Chong BF, James JA, Arriens C, Ishimori M, Wallace DJ, Liao D, Olsen NJ. Mock Recruitment for the Study of Antimalarials in an Incomplete Lupus Erythematosus Trial. Arthritis Care Res (Hoboken). 2019 Nov;71(11):1425-1429. doi: 10.1002/acr.23802. PMID 30369087
- [Background] Olsen NJ, James JA, Arriens C, Ishimori ML, Wallace DJ, Kamen DL, Chong BF, Liao D, Chinchilli VM, Karp DR. Study of Anti-Malarials in Incomplete Lupus Erythematosus (SMILE): study protocol for a randomized controlled trial. Trials. 2018 Dec 20;19(1):694. doi: 10.1186/s13063-018-3076-7. PMID 30572906
- [Derived] Porta SV, Ugarte-Gil MF, Garcia-de la Torre I, Bonfa E, Gomez-Puerta JA, Arnaud L, Cardiel MH, Alarcon GS, Pons-Estel BA, Pons-Estel G. Controversies in Systemic Lupus Erythematosus: Are We Treating Our Patients Adequately? J Clin Rheumatol. 2022 Mar 1;28(2):e651-e658. doi: 10.1097/RHU.0000000000001803. PMID 34897194

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydroxychloroquine | Placebo Oral Capsule
Started | 93 | 94
Completed | 43 | 47
Not Completed | 50 | 47
Not completed — Achieved SLE Diagnosis | 11 | 10
Not completed — Adverse Event | 1 | 1
Not completed — Pregnancy | 2 | 2
Not completed — Lost to Follow-up | 5 | 6
Not completed — Concomitant Medications | 1 | 1
Not completed — Achieved SLE and Concomitant Meds | 1 | 0
Not completed — Other | 2 | 0
Not completed — Withdrawal by Subject | 26 | 21
Not completed — Protocol Violation | 1 | 6

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is 180 patients, after excluding 7 patients due to diagnosis of SLE confirmed after delayed labs became available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine | Placebo Oral Capsule | Total
Number analyzed (Participants) | 92 | 88 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (9.75) | 33.5 (8.58) | 33.1 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 80 | 164
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 17 | 31
  Not Hispanic or Latino | 78 | 70 | 148
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 9 | 22
  White | 68 | 66 | 134
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 92 | 88 | 180
Systemic Lupus International Cooperating Clinics (SLICC) score baseline [Number; unit: Number of criteria] — SLICC scores were determined using the defined list of 17 criteria for classification of SLE. At each visit the list was reviewed and any clinical or laboratory features that satisfied a criterion were counted. This is a cumulative score, which can only increase over time. A higher score indicates more features of lupus have been found. When a score of 4 is reached, then the participant satisfies the classification criteria for SLE. This mandates removal from the trial.
  Number of criteria
    2 criteria | 62 | 56 | 118
    3 criteria | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: SLICC Score
Description: The 2012 Systemic Lupus International Collaborating Clinics classification criteria score erythematosus Minimum value = 0 Maximum value = 17 A score of 4 or greater satisfies classification for systemic lupus erythematosus.
Time Frame: Measured every 12 weeks for 96 weeks.
Population: Analysis at each timepoint includes only the number patients who were still active in the study.
Measure: Number; unit: participants
Arm/Group | Hydroxychloroquine | Placebo Oral Capsule
Number analyzed (Participants) | 92 | 88
participants
  SLICC score of 2 : baseline | 62 | 56
  SLICC score of 2 : 12 weeks: number analyzed (Participants) | 79 | 74
  SLICC score of 2 : 12 weeks | 46 | 41
  SLICC score of 2 : 24 weeks: number analyzed (Participants) | 70 | 71
  SLICC score of 2 : 24 weeks | 35 | 40
  SLICC score of 2 : 36 weeks: number analyzed (Participants) | 61 | 62
  SLICC score of 2 : 36 weeks | 31 | 34
  SLICC score of 2 : 48 weeks: number analyzed (Participants) | 56 | 55
  SLICC score of 2 : 48 weeks | 30 | 29
  SLICC score of 2 : 60 weeks: number analyzed (Participants) | 54 | 49
  SLICC score of 2 : 60 weeks | 23 | 26
  SLICC score of 2 : 72 weeks: number analyzed (Participants) | 49 | 45
  SLICC score of 2 : 72 weeks | 21 | 24
  SLICC score of 2 : 84 weeks: number analyzed (Participants) | 45 | 47
  SLICC score of 2 : 84 weeks | 21 | 22
  SLICC score of 2 : 96 weeks: number analyzed (Participants) | 45 | 50
  SLICC score of 2 : 96 weeks | 21 | 22
  SLICC score of 3 : baseline | 30 | 32
  SLICC score of 3 : 12 weeks: number analyzed (Participants) | 79 | 74
  SLICC score of 3 : 12 weeks | 33 | 31
  SLICC score of 3 : 24 weeks: number analyzed (Participants) | 70 | 71
  SLICC score of 3 : 24 weeks | 32 | 27
  SLICC score of 3 : 36 weeks: number analyzed (Participants) | 61 | 62
  SLICC score of 3 : 36 weeks | 29 | 25
  SLICC score of 3 : 48 weeks: number analyzed (Participants) | 56 | 55
  SLICC score of 3 : 48 weeks | 24 | 25
  SLICC score of 3 : 60 weeks: number analyzed (Participants) | 54 | 49
  SLICC score of 3 : 60 weeks | 28 | 23
  SLICC score of 3 : 72 weeks: number analyzed (Participants) | 49 | 45
  SLICC score of 3 : 72 weeks | 26 | 21
  SLICC score of 3 : 84 weeks: number analyzed (Participants) | 45 | 47
  SLICC score of 3 : 84 weeks | 22 | 25
  SLICC score of 3 : 96 weeks: number analyzed (Participants) | 45 | 50
  SLICC score of 3 : 96 weeks | 24 | 26
  SLICC score of 4 or more : baseline | 0 | 0
  SLICC score of 4 or more : 12 weeks: number analyzed (Participants) | 79 | 74
  SLICC score of 4 or more : 12 weeks | 0 | 2
  SLICC score of 4 or more : 24 weeks: number analyzed (Participants) | 70 | 71
  SLICC score of 4 or more : 24 weeks | 3 | 4
  SLICC score of 4 or more : 36 weeks: number analyzed (Participants) | 61 | 62
  SLICC score of 4 or more : 36 weeks | 1 | 3
  SLICC score of 4 or more : 48 weeks: number analyzed (Participants) | 56 | 55
  SLICC score of 4 or more : 48 weeks | 2 | 1
  SLICC score of 4 or more : 60 weeks: number analyzed (Participants) | 54 | 49
  SLICC score of 4 or more : 60 weeks | 3 | 0
  SLICC score of 4 or more : 72 weeks: number analyzed (Participants) | 49 | 45
  SLICC score of 4 or more : 72 weeks | 2 | 0
  SLICC score of 4 or more : 84 weeks: number analyzed (Participants) | 45 | 47
  SLICC score of 4 or more : 84 weeks | 2 | 0
  SLICC score of 4 or more : 96 weeks: number analyzed (Participants) | 45 | 50
  SLICC score of 4 or more : 96 weeks | 0 | 2
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo Oral Capsule; For the primary outcome (SLICC classification criteria count [SLICC score]), measured every 12 weeks over a 96-week period, we used an ordinal logistic regression model to compare the estimated slopes over time for the intervention (HCQ) and placebo groups. The model accounted for the ordinal and non-decreasing properties of the SLICC score. Our null hypothesis was that the intervention slope equaled the placebo slope, with a corresponding hypothesis that the slopes were not equal; Test type: Superiority; p = 0.72, Regression, Logistic

2. Secondary Outcome: Number of Subjects With Disease Progression
Description: The number of subjects who progressed from incomplete lupus to satisfaction of classification criteria for systemic lupus erythematosus using SLICC criteria.
Time Frame: Measured up to 96 weeks.
Population: Analyzed via survival method. TIme to progression, Kaplan Meier.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo Oral Capsule
Number analyzed (Participants) | 92 | 88
Participants | 12 | 12
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo Oral Capsule; Progression to SLE was defined as the number of subjects in whom a SLICC score of 4 was recorded, up to 96 weeks; Test type: Superiority; p = 0.81, Regression, Cox

3. Secondary Outcome: Number of Subjects Meeting Disease Activity Scores Defined Below
Description: Disease activity measured by the SLE Disease Activity Index Minimum score = 0 Maximum score = 105 Higher scores indicate greater activity of lupus disease
Time Frame: Measured every 12 weeks for 96 weeks.
Population: Count includes number of participants active at each visit. Groups: Score 0-1, Score 2-3, Score 4-8.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo Oral Capsule
Number analyzed (Participants) | 92 | 88
Participants
  Baseline Score 0-1 | 43 | 45
  Week 12 Score 0-1: number analyzed (Participants) | 82 | 79
  Week 12 Score 0-1 | 44 | 37
  Week 24 Score 0-1: number analyzed (Participants) | 74 | 76
  Week 24 Score 0-1 | 36 | 45
  Week 36 Score 0-1: number analyzed (Participants) | 68 | 67
  Week 36 Score 0-1 | 36 | 38
  Week 48 Score 0-1: number analyzed (Participants) | 62 | 58
  Week 48 Score 0-1 | 35 | 36
  Week 60 Score 0-1: number analyzed (Participants) | 59 | 54
  Week 60 Score 0-1 | 35 | 32
  Week 72 Score 0-1: number analyzed (Participants) | 51 | 50
  Week 72 Score 0-1 | 28 | 34
  Week 84 Score 0-1: number analyzed (Participants) | 50 | 50
  Week 84 Score 0-1 | 33 | 35
  Week 96 Score 0-1: number analyzed (Participants) | 47 | 50
  Week 96 Score 0-1 | 29 | 36
  Baseline Score 2-3 | 28 | 23
  Week 12 Score 2-3: number analyzed (Participants) | 82 | 79
  Week 12 Score 2-3 | 27 | 20
  Week 24 Score 2-3: number analyzed (Participants) | 74 | 76
  Week 24 Score 2-3 | 24 | 17
  Week 36 Score 2-3: number analyzed (Participants) | 68 | 67
  Week 36 Score 2-3 | 16 | 13
  Week 48 Score 2-3: number analyzed (Participants) | 62 | 58
  Week 48 Score 2-3 | 13 | 12
  Week 60 score 2-3: number analyzed (Participants) | 59 | 54
  Week 60 score 2-3 | 11 | 9
  Week 72 Score 2-3: number analyzed (Participants) | 51 | 50
  Week 72 Score 2-3 | 13 | 6
  Week 84 Score 2-3: number analyzed (Participants) | 50 | 50
  Week 84 Score 2-3 | 9 | 8
  Week 96 Sc ore 2-3: number analyzed (Participants) | 47 | 50
  Week 96 Sc ore 2-3 | 10 | 9
  Baseline Score 4-8 | 21 | 20
  week 12 Score 4-8: number analyzed (Participants) | 82 | 79
  week 12 Score 4-8 | 8 | 16
  Week 24 Score 4-8: number analyzed (Participants) | 74 | 76
  Week 24 Score 4-8 | 10 | 11
  Week 36 Score 4-8: number analyzed (Participants) | 68 | 67
  Week 36 Score 4-8 | 11 | 12
  Week 48 Score 4-8: number analyzed (Participants) | 62 | 58
  Week 48 Score 4-8 | 9 | 7
  Week 60 Score 4-8: number analyzed (Participants) | 59 | 54
  Week 60 Score 4-8 | 10 | 8
  Week 72 Score 4-8: number analyzed (Participants) | 51 | 50
  Week 72 Score 4-8 | 8 | 5
  Week 84 Score 4-8: number analyzed (Participants) | 50 | 50
  Week 84 Score 4-8 | 5 | 4
  Week 96 Score 4-8: number analyzed (Participants) | 47 | 50
  Week 96 Score 4-8 | 7 | 5
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo Oral Capsule; For the SLEDAI score, we combined responses to model the following groups: * Score of 0 or 1 * Score of 2 or 3 * Score of 4, 6, or 8; Test type: Superiority; p = 0.74, Regression, Logistic

4. Secondary Outcome: Count of Participants With Defined Disease Activity
Description: Disease activity measured by the Cutaneous Lupus Erythematosus Disease Activity Index Minimum score = 0 Maximum score = 70 Higher scores indicate greater cutaneous lupus activity
Time Frame: Measured every 12 weeks for 96 weeks
Population: Data are shown for number of active patients at each timepoint. CLASI activity score is measured as 0,1,2 or 3 and higher. At some timepoints, Data are Missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo Oral Capsule
Number analyzed (Participants) | 92 | 88
Participants
  Baseline: Missing data | 0 | 0
  Baseline: Score 0 | 67 | 66
  Baseline: Score 1 | 9 | 10
  Baseline: Score 2 | 8 | 9
  Baseline: Score 3 or higher | 8 | 3
  Week 12: number analyzed (Participants) | 82 | 79
  Week 12: Missing data | 4 | 6
  Week 12: Score 0 | 59 | 51
  Week 12: Score 1 | 8 | 10
  Week 12: Score 2 | 3 | 7
  Week 12: Score 3 or higher | 8 | 5
  Week 24: number analyzed (Participants) | 74 | 76
  Week 24: Missing data | 5 | 3
  Week 24: Score 0 | 52 | 61
  Week 24: Score 1 | 9 | 3
  Week 24: Score 2 | 3 | 5
  Week 24: Score 3 or higher | 5 | 4
  Week 36: number analyzed (Participants) | 68 | 67
  Week 36: Missing data | 5 | 4
  Week 36: Score 0 | 50 | 49
  Week 36: Score 1 | 5 | 4
  Week 36: Score 2 | 3 | 5
  Week 36: Score 3 or higher | 5 | 5
  Week 48: number analyzed (Participants) | 62 | 58
  Week 48: Missing data | 5 | 3
  Week 48: Score 0 | 45 | 44
  Week 48: Score 1 | 5 | 4
  Week 48: Score 2 | 2 | 2
  Week 48: Score 3 or higher | 5 | 5
  Week 60: number analyzed (Participants) | 59 | 54
  Week 60: Missing data | 3 | 5
  Week 60: Score 0 | 42 | 38
  Week 60: Score 1 | 7 | 4
  Week 60: Score 2 | 3 | 3
  Week 60: Score 3 or higher | 4 | 4
  Week 72: number analyzed (Participants) | 51 | 50
  Week 72: Missing data | 2 | 5
  Week 72: Score 0 | 42 | 40
  Week 72: Score 1 | 3 | 1
  Week 72: Score 2 | 3 | 2
  Week 72: Score 3 or higher | 1 | 2
  Week 84: number analyzed (Participants) | 50 | 50
  Week 84: Missing data | 4 | 3
  Week 84: Score 0 | 39 | 40
  Week 84: Score 1 | 2 | 1
  Week 84: Score 2 | 5 | 4
  Week 84: Score 3 or higher | 0 | 2
  Week 96: number analyzed (Participants) | 47 | 50
  Week 96: Missing data | 1 | 0
  Week 96: Score 0 | 36 | 43
  Week 96: Score 1 | 5 | 3
  Week 96: Score 2 | 4 | 2
  Week 96: Score 3 or higher | 1 | 2
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo Oral Capsule; For analysis, we combined responses ≥3 to model the following groups: * Score of 0 * Score of 1 * Score of 2 * Score of 3 or higher; Test type: Superiority; p = 0.77, Regression, Logistic; Ordinal logistic regression

5. Secondary Outcome: Patient Reported Outcome Physical Function
Description: The PROMIS 29 Adult Profile: Physical Function T Scores The T-score has a mean of 50 and a standard deviation of 10 within the reference (healthy) population.
  Higher score indicates better physical function
Time Frame: Measured every 12 weeks for 96 weeks
Population: Only patients active at each visit are measured.
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Hydroxychloroquine | Placebo Oral Capsule
Number analyzed (Participants) | 92 | 88
T score
  Baseline | 48.5 (8.26) | 48.9 (7.87)
  12 weeks: number analyzed (Participants) | 81 | 79
  12 weeks | 49.6 (7.71) | 49.7 (7.84)
  24 weeks: number analyzed (Participants) | 72 | 75
  24 weeks | 49.5 (7.73) | 49.4 (8.42)
  36 weeks: number analyzed (Participants) | 65 | 65
  36 weeks | 48.8 (8.12) | 49.2 (8.6)
  48 weeks: number analyzed (Participants) | 59 | 58
  48 weeks | 48.6 (8.3) | 49.9 (7.89)
  60 weeks: number analyzed (Participants) | 59 | 54
  60 weeks | 49.6 (8.06) | 49.4 (7.92)
  72 weeks: number analyzed (Participants) | 51 | 50
  72 weeks | 49.3 (8.28) | 50.1 (8.24)
  84 weeks: number analyzed (Participants) | 47 | 50
  84 weeks | 49.7 (7.84) | 48.7 (8.55)
  96 weeks: number analyzed (Participants) | 46 | 50
  96 weeks | 48.5 (8.17) | 50.1 (7.93)
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo Oral Capsule; Test type: Superiority; p = 0.386, t-test, 2 sided; Paired t-test

6. Secondary Outcome: Patient Reported Outcomes Fatigue
Description: Selected Patient-reported outcomes measurement information system (PROMIS) fatigue items T Scores are reported. The T-score has a mean of 50 and a standard deviation of 10 within the reference (healthy) population.
  Higher scores indicate more fatigue
Time Frame: Measured every 12 weeks for up to 96 weeks
Population: Only active patients are recorded at each visit. Values represent Fatigue T-scores.
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Hydroxychloroquine | Placebo Oral Capsule
Number analyzed (Participants) | 92 | 88
T score
  Baseline: number analyzed (Participants) | 91 | 79
  Baseline | 54.7 (10.8) | 55.0 (10.87)
  12 weeks: number analyzed (Participants) | 82 | 77
  12 weeks | 53.0 (10.6) | 53.1 (11.2)
  24 weeks: number analyzed (Participants) | 72 | 75
  24 weeks | 52.2 (10.2) | 53.2 (12.0)
  36 weeks: number analyzed (Participants) | 64 | 66
  36 weeks | 52.3 (10.5) | 51.8 (11.4)
  48 weeks: number analyzed (Participants) | 60 | 58
  48 weeks | 51.5 (10.6) | 51.4 (11.3)
  60 weeks: number analyzed (Participants) | 58 | 51
  60 weeks | 51.1 (11.0) | 49.1 (9.8)
  72 weeks: number analyzed (Participants) | 51 | 50
  72 weeks | 50.9 (11.2) | 50.3 (11.2)
  84 weeks: number analyzed (Participants) | 47 | 50
  84 weeks | 51.7 (8.6) | 51.1 (10.5)
  96 weeks: number analyzed (Participants) | 46 | 50
  96 weeks | 51.9 (11.3) | 50.7 (11.0)
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo Oral Capsule; Test type: Superiority; p = 0.497, t-test, 2 sided; Paired t-test

7. Secondary Outcome: Physician Global Asssessment
Description: Physician Global Visual Analogue Scale Minimum score = 0 Maximum score = 1.0 Higher scores indicate worse status
Time Frame: Measured every 12 weeks for up to 96 weeks
Population: Number of active patients at each time point are measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo Oral Capsule
Number analyzed (Participants) | 92 | 88
Participants
  Baseline: Missing data | 1 | 1
  Baseline: Score 0 | 39 | 40
  Baseline: Score 0.25 | 35 | 31
  Baseline: Score 0.50 | 14 | 14
  Baseline: Score 0.75 or higher | 3 | 2
  Week 12: number analyzed (Participants) | 82 | 79
  Week 12: Missing data | 4 | 7
  Week 12: Score 0 | 46 | 39
  Week 12: Score 0.25 | 23 | 23
  Week 12: Score 0.50 | 4 | 8
  Week 12: Score 0.75 or higher | 5 | 2
  Week 24: number analyzed (Participants) | 74 | 76
  Week 24: Missing data | 4 | 4
  Week 24: Score 0 | 35 | 43
  Week 24: Score 0.25 | 24 | 19
  Week 24: Score 0.50 | 9 | 7
  Week 24: Score 0.75 or higher | 2 | 3
  Week 36: number analyzed (Participants) | 68 | 67
  Week 36: Missing data | 6 | 6
  Week 36: Score 0 | 41 | 34
  Week 36: Score 0.25 | 15 | 16
  Week 36: Score 0.50 | 5 | 7
  Week 36: Score 0.75 or higher | 1 | 4
  Week 48: number analyzed (Participants) | 62 | 58
  Week 48: Missing data | 5 | 3
  Week 48: Score 0 | 39 | 37
  Week 48: Score 0.25 | 14 | 11
  Week 48: Score 0.50 | 4 | 5
  Week 48: Score 0.75 or higher | 0 | 2
  Week 60: number analyzed (Participants) | 59 | 54
  Week 60: Missing data | 4 | 6
  Week 60: Score 0 | 33 | 33
  Week 60: Score 0.25 | 13 | 6
  Week 60: Score 0.50 | 7 | 7
  Week 60: Score 0.75 or higher | 2 | 2
  Week 72: number analyzed (Participants) | 51 | 50
  Week 72: Missing data | 4 | 5
  Week 72: Score 0 | 25 | 29
  Week 72: Score 0.25 | 19 | 15
  Week 72: Score 0.50 | 3 | 1
  Week 72: Score 0.75 or higher | 0 | 0
  Week 84: number analyzed (Participants) | 50 | 50
  Week 84: Missing data | 4 | 3
  Week 84: Score 0 | 35 | 37
  Week 84: Score 0.25 | 8 | 9
  Week 84: Score 0.50 | 3 | 1
  Week 84: Score 0.75 or higher | 0 | 0
  Week 96: number analyzed (Participants) | 47 | 50
  Week 96: Missing data | 2 | 1
  Week 96: Score 0 | 31 | 38
  Week 96: Score 0.25 | 11 | 6
  Week 96: Score 0.50 | 2 | 3
  Week 96: Score 0.75 or higher | 1 | 2
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo Oral Capsule; Test type: Superiority; p = 0.99, Regression, Logistic; Ordinal logistic regression

8. Secondary Outcome: Fluorescence Intensity (FI) of Autoantibodies in Serum
Description: Fluorescence intensity of Autoantibodies will be measured using a slide array. Minimum score is 0.1 Maximum score >100 A higher score indicates higher level of the autoantibody being measured.
Time Frame: Measured at baseline and final visit up to 96 weeks.
Population: Only patients who completed or who had a defined final visit are included. Samples were measured at baseline and last visit.
Measure: Mean (Standard Deviation); unit: Mean Fluorescence Intensity
Arm/Group | Hydroxychloroquine | Placebo Oral Capsule
Number analyzed (Participants) | 74 | 78
Mean Fluorescence Intensity
  Baseline CENP-A | 1319 (869) | 1243 (1222)
  Baseline CENP-B | 5461 (2703) | 5454 (3029)
  Baseline dsDNA | 2838 (2766) | 2582 (4289)
  Baseline Genomic DNA | 4484 (7821) | 3362 (2458)
  Baseline HIstone | 2349 (2118) | 2145 (1703)
  Baseline IFN-alpha | 1813 (1619) | 2049 (1960)
  Baseline IFN-gamma | 9092 (6184) | 9373 (7330)
  Baseline IL-17A | 9991 (6075) | 9953 (5816)
  Baseline KU. (P70/P80) | 3933 (5283) | 3967 (5697)
  Baseline La/SSB | 4682 (9508) | 4703 (10076)
  Baseline Laminin | 16234 (17545) | 15573 (16455)
  Baseline Liver Baseline Cytosol ' | 3563 (3632) | 3267 (3074)
  baseline LKM 1 | 3067 (1321) | 2903 (1151)
  Baseline MDA5 | 3725 (4064) | 3483 (3476)
  Baseline Mi-2 | 1140 (760) | 1067 (679)
  Baseline NRP1 | 23735 (20781) | 24296 (21025)
  Baseline Nucleolin | 3108 (2148) | 2748 (1576)
  Baseline Nucleosome | 3017 (1661) | 2800 (1255)
  Baseline NXP2 | 3765 (2275) | 3584 (2228)
  Baseline PL-7 | 2681 (1335) | 2352 (973)
  Baseline PL-12 | 6040 (2533) | 5672 (1905)
  Baseline PM/SCL-100 | 2967 (2631) | 2650 (1919)
  Baseline Ro/SSA 60 KDA | 1800 (4705) | 1879 (5617)
  Baseline Scl-70 | 1596 (1499) | 1569 (1231)
  Baseline Sm | 1347 (1677) | 1135 (1087)
  Baseline thyroglobulin | 4211 (7237) | 2933 (4782)
  Baseline TPO | 7986 (9281) | 6769 (7279)
  Baseline tTG | 6966 (4280) | 6381 (3164)
  Baseline U1-snRNPA | 2372 (2869) | 2184 (2701)
  Baseline U1-snRNP C | 657 (819) | 602 (821)
  Baseline U1-snRNP B/B | 260 (110) | 252 (94)
  Baseline Vimentin | 3160 (1670) | 3006 (1140)
  Final CENP-A | 1243 (1222) | 1889 (7462)
  Final CENP-B | 5454 (3029) | 6367 (8328)
  Final dsDNA | 2582 (4289) | 2496 (2472)
  Final Genomic DNA | 3362 (2458) | 3595 (3971)
  Final Histone | 2145 (1703) | 2304 (2636)
  Final IFN-alpha | 2049 (1960) | 2150 (2096)
  Final IFN-gamma | 9373 (7330) | 10235 (6071)
  Final IL-17A | 9953 (5816) | 11656 (6798)
  Final Ku P70/P80 | 3967 (5697) | 4209 (4440)
  Final La/SS-B | 4703 (10076) | 2881 (1677)
  Final Laminin | 15573 (16455) | 18192 (19262)
  Final Liver Cytosol 1 | 3267 (3074) | 3538 (3506)
  Final LKM 1 | 2903 (1151) | 3323 (1549)
  Final MDA5 | 3483 (3476) | 4262 (2636)
  Final Mi-2 | 1067 (679) | 1299 (736)
  Final Nrp1 | 24296 (21025) | 25597 (22237)
  Final Nucleolin | 2748 (1576) | 3721 (2291)
  Final Nucleosome | 2800 (1255) | 3292 (1595)
  Final NXP2 | 3584 (2228) | 4598 (2627)
  Final PL-7 | 2352 (973) | 2861 (1790)
  Final PL-12 | 5672 (1905) | 6673 (2873)
  Final PM/Scl 100 | 2650 (1919) | 2982 (1768)
  Final Ro/SS-A 60 Kda | 1879 (5617) | 1421 (908)
  Final Scl-70 | 1569 (1231) | 2009 (4108)
  Final Sm | 1135 (1087) | 1858 (5755)
  Final Thyroglobulin | 2933 (4782) | 3651 (6602)
  Final TPO | 6769 (7279) | 6873 (4793)
  Final tTg | 6381 (3164) | 6356 (2314)
  Final U1-snRNP A | 2184 (2701) | 2845 (7385)
  Final U1-snRNP C | 657 (819) | 502 (276)
  Final U1-snRNP B/B | 260 (110) | 247 (92)
  Final Vimentin | 3160 (1670) | 3891 (1542)
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo Oral Capsule; Test type: Superiority; p > 0.05, t-test, 2 sided

9. Secondary Outcome: Ophthalmologic Toxicity as Measured by Snellen Visual Acuity
Description: Snellen visual acuity measured in right and left eyes Scale 10 to 50 with higher numbers indicating lower visual acuity Number of participants with each level of visual acuity in right eye and left eye are counted in the two groups at the final visit
Time Frame: Measured at up to 96 weeks or final visit
Population: Only patients who completed the exams are analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo Oral Capsule
Number analyzed (Participants) | 52 | 55
Participants
  Right Eye: Missing data | 6 | 7
  Right Eye: 10 | 0 | 0
  Right Eye: 15 | 4 | 6
  Right Eye: 20 | 34 | 36
  Right Eye: 25 | 6 | 5
  Right Eye: 30 | 2 | 1
  Right Eye: 50 | 0 | 0
  Left eye: Missing data | 6 | 7
  Left eye: 10 | 1 | 0
  Left eye: 15 | 4 | 6
  Left eye: 20 | 33 | 38
  Left eye: 25 | 7 | 2
  Left eye: 30 | 1 | 1
  Left eye: 50 | 0 | 1
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo Oral Capsule; Test type: Non-Inferiority — Outcome with hydroxychloroquine is hypothesized to be not inferior to outcome with placebo; p > 0.5, Fisher Exact

10. Secondary Outcome: Ophthalmologic Toxicity by Humphrey Visual Field Testing
Description: Number of participants with abnormal visual field testing at the final visit.
Time Frame: Measured at final visit up to 96 weeks
Population: only patients who completed the exams are shown.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo Oral Capsule
Number analyzed (Participants) | 52 | 55
Participants | 0 | 0
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo Oral Capsule; Test type: Superiority; p = 1.00, Fisher Exact

11. Secondary Outcome: Ophthalmologic Toxicity as Measured by Spectral Domain Ocular Coherence Tomography.
Description: Number of participants with abnormal spectral domain ocular coherence tomography at final visit
Time Frame: Measured at up to 96 weeks or final visit
Population: only patients who completed exams are shown
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo Oral Capsule
Number analyzed (Participants) | 52 | 55
Participants | 0 | 0
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo Oral Capsule; Test type: Superiority; p = 1.00, Fisher Exact

ADVERSE EVENTS:
Time Frame: Up to 96 weeks.
Arm/Group | Hydroxychloroquine | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/88
Serious Adverse Events (participants affected / at risk) | 4/92 | 5/88
Other Adverse Events (participants affected / at risk) | 83/92 | 85/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=92) | Placebo Oral Capsule (N=88)
Hospitalization Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Colitis
Hospitalization Uterine Fibroids (Reproductive system and breast disorders) | 0 | 1 (1) — Uterine Fibroids
Hospitalization Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) — Peripheral sensory neuropathy
Hospitalization COVID-19 (Infections and infestations) | 0 (0) | 1 (1) — COVID-19 infection
Hospitalization Thromboembolic event (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hospitalization Cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hospitalization Radiculitis (Nervous system disorders) | 0 (0) | 1 (1)
Hospitalization Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Hospitalization Mastectomy (Surgical and medical procedures) | 1 (1) | 0 (0) — Right mastectomy, benign
Hospitalization Bilateral capsulotomy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=92) | Placebo Oral Capsule (N=88)
Upper Respiratory Infection (Infections and infestations) | 11 (11) | 11 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 11 (11)
Flu like symptoms (Infections and infestations) | 9 (9) | 7 (7)
Headache (Nervous system disorders) | 9 (9) | 7 (7)
COVID-19 Infection (Infections and infestations) | 7 (7) | 9 (9)
Nausea (Gastrointestinal disorders) | 8 (8) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (6) — Maculo-papular rash
Urinary Tract Infection (Infections and infestations) | 5 (5) | 6 (6)
Dry Skin (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5)
Sinusitis (Infections and infestations) | 6 (6) | 4 (4)
Vaginal infection (Reproductive system and breast disorders) | 5 (5) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)

LIMITATIONS AND CAVEATS:
The number of participants was lower than planned in part due to the restrictions that were in place during the COVID-19 pandemic; some sites were closed for a time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT03030118/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT03030118/ICF_001.pdf